CLINICAL TRIAL: NCT06453577
Title: Pharmacokinetics and Pharmacodynamics of Bisoprolol and SGLT2-Inhibitors (Dapagliflozin, Empagliflozin) in Acutely Decompensated Heart Failure BISO-ADHF (BI=BIsoprolol, SO=Sodium-glucose Co-transporter-2 Inhibitors in Acute Decompensated Heart Failure)
Brief Title: Pharmacokinetics of Bisoprolol and SGLT2i in Acutely Decompensated Heart Failure
Acronym: BISO-ADHF
Status: Active, not recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: BISO-ADHF
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute Decompensated Heart Failure; Bisoprolol; SGLT2-inhibitors; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with acute decompensated heart failure: Patients presenting with acute decompensated heart failure (ADHF) at Saarland University Medical Center. (phase A)
  ADHF (acutely decompensated CHF or new onset/ de novo HF):
  Evidence of congestion and decompensation defined by physical abnormalities as follows: Physical evidence of congestion, including pitting edema > 2 mm in the lower extremities extending from the ankles to mid-calf and rales on pulmonary examination (chest X-ray)
  Interventions: Drug: Recompensation (guideline directed medical therapy)
- Patients after recompensation: Same patients after recompensation. (phase B)
  After resolution of the signs of congestion (mainly achieved by intravenous diuretics and/or vasodilators but no requirement for positive inotropic drugs such as catecholamines or levosimendan), as evidenced by the following:
  1. A decrease in body weight and
  2. Resolution of the physical findings (absence of signs) of congestion, including resolution of the physical findings of congestion including peripheral edema and rales on pulmonary examination (chest X-ray) according to the clinical judgment of the attending physician.

INTERVENTIONS:
Drug: Recompensation (guideline directed medical therapy) — Recompensation mainly achieved by intravenous diuretics and/or vasodilators but no requirement for positive inotropic drugs such as catecholamines or levosimendan.
  Groups: Patients with acute decompensated heart failure

SUMMARY:
The pharmacokinetics (PK) and pharmacodynamics (PD) of bisoprolol and sodium-glucose co-transporter-2 inhibitors (SGLT2i, dapagliflozin and empagliflozin) in patients with acutely decompensated heart failure (ADHF), compared to the recompensated state, is unknown. If not in cardiogenic shock (no need of vasopressor (catechoalmines) therapy or other inotropic support), established oral betablocker therapy should de continued. Whether this holds true for SGLT2i in ADHF is less clear but current evidence suggest safety and potentially beneficial effects in doing so.

To the best of our knowledge, no data regarding PK/PD are available for the most widely used beta blocker bisoprolol and the newly approved/in Germany available SGLT2i Dapagliflozin and Empagliflozin. This study shall provide first evidence on the PK/PD-profile of p.o. bisoprolol and SGLT2i (dapaglifozin or empagliflozin) regarding acute (hemodynamic) effects and safety as well as to provide data on dose recommendations eventually in patients with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with decompensated heart failure caused by heart failure irrespective of ejection fraction (heart failure with reduced, mildly reduced or preserved ejection fraction and de-novo heart failure)
* Signs of decompensation: peripheral edema, jugular venous distension, pulmonary rales, protodiastolic gallop rhythm, ascites, or demonstration of pulmonary venous congestion on chest X-ray
* Previous documented beta blocker therapy
* elevated natriuretic peptides (nt-pro-BNP ≥125 pg/ml)
* patients admitted to the intensive care unit

Exclusion Criteria:

* Left ventricular or biventricular assist device therapy
* Cardiogenic shock
* need of vasopressor (catechoalmines) therapy or other inotropic support (dobutamine or levosimendan)
* Clinical symptomatic hypotension
* Bradycardia (<50 bpm)
* patients requiring dialysis (CVVHD)
* Inflammatory bowel disease (eg, M. Crohn or Colitis ulcerosa)
* Not able to give written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute decompensated heart failure (ADHF) at the intensive care unit at Saarland University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax in ng/ml] of Bisoprolol/ Dapagliflozin/ Empaglifozin | up to 7 days
  toxicological measurements (using liquid chromatography coupled to high-resolution mass spectrometry) of drug levels in venous blood in decompensated and recompensated state (Comparison decompensated and recompensated state)
Plasma Concentration (in ng/ml) over time of Bisoprolol/ Dapaglifozin/ Empagliflozin (AUC= Area under the curve) | up to 7 days
  toxicological measurements (using liquid chromatography coupled to high-resolution mass spectrometry) of drug levels in venous blood in decompensated and recompensated state (Comparison decompensated and recompensated state)

SECONDARY OUTCOMES:
Hemodynamic assessment (blood pressure in mmHg) of patients in decompensated and recompensated state | up to 7 days
  Pharmacodynamics of Bisoprolol and Dapagliflozin and Empagliflozin
Hemodynamic assessment (heart rate in bpm) of patients in decompensated and recompensated state | up to 7 days
  Pharmacodynamics of Bisoprolol and Dapagliflozin and Empagliflozin

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine III, Cardiology, Angiology and Intensive Care Medicine, University Hospital Saarland, Saarland University, Homburg, Germany

IPD SHARING:
Plan to Share IPD: No